CLINICAL TRIAL: NCT00767858
Title: Cultural Congruence in International Genetics Research: Perceptions of Opportunities and Challenges Among Researchers
Brief Title: Cultural Congruence in International Genetics Research
Status: Terminated | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999908225; 08-HG-N225
Record Dates: First submitted 2008-10-06; First posted 2008-10-07 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2016-02-24

CONDITIONS: Cultural Diversity
Keywords: Genetic; Genetic Literacy; Human Genetic Research; Cultural Congruence; Interview

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
This study will explore how cultural differences influence genetics research in developing countries. Human genetics research is becoming more common in developing countries. However, when research is conducted with people living in developing countries, there is a chance that culture differences can lead to misunderstandings between investigators and participants, resulting in ineffective research. This study will explore challenges facing investigators conducting genetics research in developing countries and opportunities to improve this kind of research.

Scientists who have conducted genetics research in a developing country may be eligible to participate in this study. Participants are interviewed by telephone. The interview, which lasts about an hour, includes questions about the researchers decision to conduct the study they have done, the times they noticed that culture played a role in the research and the times that were more challenging and less challenging.

The interviews are recorded, transcribed and analyzed for themes related to cultural congruence and specific challenges and opportunities with regard to cultural congruence.

DETAILED DESCRIPTION:
The objective of the proposed study is to describe cultural congruence, including diversity, awareness, sensitivity, and competence in people conducting human genetics research in developing countries, as well as to explore challenges and opportunities to improve cultural congruence. Human genetics research is becoming more common in developing countries, as researchers take advantage of differences in environment and population diversity. However, when research is conducted with individuals living in developing countries, there is a chance that culture will lead to misunderstandings between investigators and participants and consequently ineffective research. The proposed study uses a cross-sectional semi-structured qualitative interview design. Thirty to forty-five participants will be recruited. Participants will be researchers with experience in conducting genetics research in developing countries, who will have had direct contact with the participants in their research studies. These researchers will be recruited from professional organizations, through identification of lead authors in literature searches, and through snowball recruitment. Interviews will be conducted by telephone, recorded, transcribed, and analyzed for themes related to cultural congruence and specific challenges and opportunities with regard to cultural congruence.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Participants will include genetics researchers who have had direct contact with participants in human genetic research in developing countries. A researcher may be defined as any project staff, faculty, or investigator involved in carrying out a genetics research protocol in a developing country. Project staff are included as potential participants so that whoever has most contact with genetic research participants is able to participate in the proposed study.
* Researchers will be able to decide whether the country that they are working in is defined as a developing country, as opposed to dictating a fixed list of countries that qualify. This will be assessed by participant report during the screening process.

EXCLUSION CRITERIA:

* Researchers who do research in developing countries but do not have direct contact with human participants.
* Participants who are non-English-speaking or under the age of 18.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2008-09-24; Study Completion 2016-02-24

CONTACTS AND LOCATIONS:
Overall Officials: Barbara B Biesecker, Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (1):
- National Human Genome Research Institute (NHGRI), 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Betancourt JR, Green AR, Carrillo JE, Ananeh-Firempong O 2nd. Defining cultural competence: a practical framework for addressing racial/ethnic disparities in health and health care. Public Health Rep. 2003 Jul-Aug;118(4):293-302. doi: 10.1093/phr/118.4.293. PMID 12815076
- [Background] Ezeome ER, Marshall PA. Informed consent practices in Nigeria. Dev World Bioeth. 2009 Dec;9(3):138-48. doi: 10.1111/j.1471-8847.2008.00234.x. Epub 2008 Apr 29. PMID 18452553
- [Background] Chokshi DA, Thera MA, Parker M, Diakite M, Makani J, Kwiatkowski DP, Doumbo OK. Valid consent for genomic epidemiology in developing countries. PLoS Med. 2007 Apr;4(4):e95. doi: 10.1371/journal.pmed.0040095. PMID 17455985